CLINICAL TRIAL: NCT00185354
Title: Multi-center, Open, Randomized, Parallel Group Comparison of Cycle Control for Seven Cycles and Endometrial Safety in a Subgroup for Thirteen Cycles of Contraceptive Patch SH P00331F (0.9 mg Ethinylestradiol/1.9 mg Gestodene) vs. a Contraceptive Comparator Patch (0.6 mg Ethinylestradiol/6 mg Norelgestromin) in 400 Healthy Female Volunteers
Brief Title: FC Patch Comparator Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91402; 2004-000821-31 (EudraCT Number); 307969 (Other: Study Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Contraception
Keywords: FC patch; comparator study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-5016, SH P00331F
- Arm 2 (Active Comparator)
  Interventions: Drug: SH P00331N

INTERVENTIONS:
Drug: BAY86-5016, SH P00331F — Drug amount per patch: 0.9 mg EE2 + 1.9 mg gestodene (GSD)
  Arms: Arm 1
Drug: SH P00331N — Drug amount per patch: 0.6 mg EE2 + 6 mg NGM
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare bleeding pattern and safety of contraceptive patch SH P00331F to a marketed comparator.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer aged 18-35, smokers 18-30

Exclusion Criteria:

* Contraindications for using hormonal contraceptives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2004-11; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Bleeding pattern and cycle control | 13 cycles
Number of pregnancies | 13 cycles

SECONDARY OUTCOMES:
Adverse events collection | 13 cycles
Endometrial biopsy | 13 cycles
Physical and gynecological exam | 13 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (24):
- Austria (5):
  - Wörgl, Tyrol
  - Bregenz
  - Graz
  - Vienna
  - Zeltweg
- Finland (2):
  - Helsinki
  - Turku
- France (11):
  - Paris, Paris
  - Biarritz
  - Bordeaux
  - Compiègne
  - Maisons Lafitte
  - Montargis
  - Nancy
  - Pantin
  - Roanne
  - Saint-Germain-en-Laye
  - Toulouse
- Spain (6):
  - San Fernando, Cádiz
  - Pontevedra, Galicia
  - Salt, Girona
  - Guadalajara, Guadalajara
  - Barcelona
  - Santiago de Compostela

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/